CLINICAL TRIAL: NCT06593418
Title: A Phase I/II Study of Cardiac Radioablation for Refractory Ventricular Tachycardia
Brief Title: Cardiac Radioablation for VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, John Robertson, MD, Clinical Director, Radiation Oncology, Corewell Health East
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-069
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Ventricular Tachycardia; Myocardial Infarction
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Infarction | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Radiation Therapy at 15 Gy for Ventricular Tachycardia (Experimental): Post myocardial infarction patients with refractory ventricular tachycardia requiring cardio ablation, treated with 15 Gy
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Radiation Therapy at 20 Gy for Ventricular Tachycardia (Experimental): Post myocardial infarction patients with refractory ventricular tachycardia requiring cardio ablation, treated with 20 Gy
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Radiation Therapy at 25 Gy for Ventricular Tachycardia (Experimental): Post myocardial infarction patients with refractory ventricular tachycardia requiring cardio ablation, treated with 25 Gy
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Stereotactic body radiation therapy, which delivers precise, high-dose radiation non-invasively to generate thermal scarring to myocardial targets causing VT

SUMMARY:
The goal of this interventional study is to determine the minimum dose necessary for successful cardiac radioablation of refractory ventricular tachycardia (VT) and to study the utility of target volume definition using Delayed Enhancement Cardiac MRI (DE-CMR) .

DETAILED DESCRIPTION:
This voluntary study is designed to learn what is the minimum dose of radiation therapy (RT) needed to successfully reduce the incidence of refractory ventricular tachycardia (VT) by half. Additionally, the study will examine the utility of target volume definition using Delayed Enhancement Cardiac MRI (DE-CMR). Radiation therapy, given in a highly focused single dose to a portion of the heart, by a non-invasive method, has been found to change the electrical conduction of the heart. This will be done with the goal of reducing the number of episodes of VT in people where invasive thermal (heat) ablation and heart medications have not completely worked.

Cardiac radioablation has been done at other institutions using a dose of RT that may be higher than needed to obtain the benefit of fewer episodes of VT. We are trying to learn if lower doses of RT will work to reduce VT. Cardiac radioablation is currently offered at a number of institutions worldwide at the standard dose of 25 Gray, or Gy (the unit of dose for radiation therapy) given in a single treatment. This study is testing if lower doses of RT are just as effective as 25 Gy. The doses being tested are 15 Gy (the dose that we will start at), 20 Gy and 25 Gy (if the lower doses are found not to work well).

Potential participants will be identified by their cardiologist. Electroanatomic mapping will have already been obtained as part of routine care. A Delayed Enhancement Cardiac MRI will be performed (if a new one is necessary) and a Radiation Therapy Simulation. Commercial RT software will be used to fuse the DE CMR and the RT Simulation treatment planning CT scan. The cardiologist and radiation oncologist will define the Gross Target Volume and the expansions for the Clinical and Planning Target Volumes. These volume definitions will be used by the Radiation Oncology Dosimetrist. The dose will be determined in standard 3+3 Phase I fashion. Dose escalation will proceed in a standard 3 + 3 Phase I fashion according to both dose limiting toxicity (DLT) and efficacy. Escalation will stop when there is efficacy 50% or greater without severe DLT or when there is severe DLT (2+ of 3 or 6 with DLT as per traditional 3 + 3 Phase I design). The dose will not be escalated within a single patient.

When the minimum effective dose (MED) or maximum tolerable dose (MTD) is determined, further accrual will occur at that dose level until 12 patients are accrued and observed for 14 weeks (6 week blanking and 8 week (56 day) evaluation).

DLT is defined as any grade 3 toxicity requiring hospitalization or any grade 4 - 5 toxicity (CTCAE v.5) determined to be treatment related (possibly, probably, or definitely related to study treatment) occurring within 14 weeks after treatment. DLT's occurring after the 14-week observation period may still impact on dose escalation.

Efficacy is defined as a 50% or higher reduction in the number of episodes of VT archived over the 56 days before treatment (obtained from their automatic internal cardiac defibrillator (AICD) device) versus over a consecutive 56 days after treatment starting after the 6-week post-treatment blanking period.

Treatment will be given using standard SBRT technique. The week 14 assessment will be used to determine efficacy (defined as a 50% of higher reduction in the number of episodes of VT archived over the 56 days before treatment versus over a consecutive 56 days after treatment starting after the 6 week post-treatment blanking period).

Following determination of the study dose in the Phase I portion of the study, a Phase II portion will be performed until a total of 12 patients are accrued at the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older.
* Automatic implanted cardiac defibrillator present.
* VT is monomorphic with at least two episodes of VT within an eight week (56 day) period as recorded by an AICD or heart failure related to VT or VT storm.
* Ejection fraction ≥20%.
* At least one previous cardiac ablation for VT.
* VT refractory despite antiarrhythmic medications.
* Likely to live for 12 months in the absence of VT.
* AICD in a position in the chest RT to be given without direct radiation.
* Woman of reproductive age must ensure that she won't become pregnant or breastfeed at the time of RT.
* The participant has no contraindications to a Cardiac MRI as per routine Cardiology practice.

Exclusion Criteria:

* Class IV heart failure
* Abandoned leads.
* Prior radiation therapy to the chest or upper abdomen.
* Interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in number of ventricular tachycardia (VT) episodes from pre-cardiac radioablation to post-cardiac radioablation | 56 days pre-treatment and 98 days post treatment (42 day blanking period plus 56 days)
  Change in the number of episodes of VT over the 56 days before treatment versus over a consecutive 56 days post treatment (following the 6 week post-treatment blanking period). A negative number represents a reduction in episodes after treatment (improved function) and a positive number represents an increase in episodes after treatment (worsened function).
Dose limiting toxicity | 14 weeks
  Number of participants who had dose limiting toxicity defined as any grade 3 toxicity requiring hospitalization or any grade 4-5 toxicity determined to be treatment-related.

SECONDARY OUTCOMES:
Efficacy of ablation using target volume definition with Delayed Enhancement Cardiac MRI (DE-CMR) | 56 days pre-treatment and 98 days post treatment (42 day blanking period plus 56 days)
  Number of participants who had successful cardiac radioablation using target volume definition DE-CMR, defined as a 50% or higher reduction in the number of episodes of VT archived over the 56 days before treatment (obtained from their automatic internal cardiac defibrillator (AICD) device) versus over a consecutive 56 days after treatment starting after the 6-week post-treatment blanking period.

CONTACTS AND LOCATIONS:
Overall Officials: John Robertson, MD, Principal Investigator — Corewell Health William Beaumont University Hospital
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No